CLINICAL TRIAL: NCT07116408
Title: Intranasal Sphenopalatine Ganglion Blockade as a Non-invasive, Opioid-sparing Treatment for Headaches Following Aneurysmal Subarachnoid Hemorrhage
Brief Title: Intranasal Sphenopalatine Ganglion Blockade for Headaches Following Aneurysmal Subarachnoid Hemorrhage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Principal Investigator, John Terry, Associate professor of Neurology, Wright State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-196
Record Dates: First submitted 2025-06-18; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage (aSAH); Headache
Keywords: Headache; subarachnoid hemorrhage; aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache; Aneurysm | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Treatment arm
  Interventions: Drug: Lidocaine (drug); Device: Tx 360

INTERVENTIONS:
Drug: Lidocaine (drug) — Tx 360/lidocaine
Device: Tx 360 — Tx 360 device

SUMMARY:
In patients with bleeding from a brain aneurysm, severe headache is the most common complaint. However, the pain is difficult to treat. The use of standard pain medications is common, but pain control remains poor. Additionally, pain medicines have multiple side effects including sedation, interference with breathing, intestinal cramping, low blood pressure, and the risk of addiction. In the present study, the investigators will examine the use of a medication to block the sphenopalatine ganglion which is a bundle of nerves that includes nerves that cause head pain. This block is performed by spraying numbing medication into the back of the nasal cavity on both sides. This particular pain medication does not have the side effects discussed above. The purpose of the study is to see if this treatment will decrease pain without causing unwanted side effects.

All patients in the study will receive standard pain medicine as needed for headache. Information will be collected from the patient's medical chart on the amount of pain medication used and the amount of pain the patient describes having. The average pain will be calculated for the first 24 hours the patient is in the hospital. At that point, the patient will receive pain medication sprayed into the back of the nasal cavity on both sides. Patients will also receive this treatment 3 days later. Following these treatments, information will be obtained on the average amount of pain, and how much other pain medication is used.

The investigators will look at the amount of pain and the amount of other pain medicine used over the first 24 hours before the nasal pain medicine treatment and compare it to the time after the treatments to see if the amount of pain decreases and if the amount of other pain medicine needed decreases as well. Six months after discharge, the patient will be contacted by phone to find out more information about how much head pain they had after discharge from the hospital.

DETAILED DESCRIPTION:
Spontaneous subarachnoid hemorrhage (SAH) accounts for up to 8% of strokes and affects approximately 30,000 individuals yearly in the US alone. Of those, ruptured intracranial aneurysm is the etiology up to 85% of the time. In these patients, severe headache is the most common complaint and its treatment is difficult and often inadequate. However, adequate. Opioids, often in escalating doses, are guideline recommended, but unfortunately they have significant side effects and are often not effective. There have been numerous trials looking at different treatments for the headache caused by SAH. There is an urgent need for an effective treatment with tolerable side effects. The pathophysiology of pain in aneurysmal subarachnoid hemorrhage (aSAH) is not well elucidated.

It is likely related to vasoactive and inflammatory byproducts of blood degradation in the subarachnoid space. The intracranial vessels themselves are abundantly innervated, predominantly by branches of the maxillary nerve. The sphenopalatine ganglion (SPG) is a possible target for intervention, as blockade has been shown to be effective in cluster headaches. The SPG is located near the maxillary nerve, which may explain why blockade is also useful in several other head pain disorders. A small, single center pilot study of seven patients evaluated a bilateral suprazygomatic pterygopalatine fossa blockade as a treatment for headache, and all the patients had clinically significant reductions in reported pain. This study aims to evaluate whether intranasal SPG blockade could provide an effective and minimally invasive treatment option to improve pain and possibly reduce opioid requirements in these patients.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 18 years or older who are being treated in the neurologic ICU for subarachnoid hemorrhage with Hunt and Hess scale of 0-3 (Scale ranges from 0 to 5 with higher numbers indicating more severe symptoms) and able to verbally report headache will be considered for inclusion in this study.

Exclusion Criteria:

* Patients under the age of 18 years of age.
* Patients with an allergy to lidocaine.
* Patients from all vulnerable groups.
* Patients with Hunt and Hess scale score of 4-5. (Scale ranges from 0 to 5 with higher numbers indicating more severe symptoms.)
* Patients who are not able to consent.
* Mentally impaired patients that are unable to provide consent.
* Patients that are prisoners.
* Pregnant patients.

Additionally, patients with contraindications to use of the Tx 360 device will be excluded. Contraindications include:

* History of recurrent nose bleeds.
* Nasal septal deformity such as cleft lip and palate, choanal atresia (narrowed nasal passages), atrophic rhinitis, rhinitis medicamentosa, septal perforation, nasal/midface trauma.
* Recent nasal/sinus surgery
* Presence of a bleeding disorder (eg., Von Willebrand's disease or hemophilia).
* Severe respiratory distress.
* Presence of angiofibroma, sinus tumor, or granulomatous disease of the nasopharynx.
* Presence of nasal trauma.
* Nasal congestion that has been present more than 10 days, high fever, or abnormal appearance of the nasal mucosa or mucus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Headache severity | Day 1 (day of consent) Patient receives first treatment. Pain will be recorded every 8 hours. Second treatment is on day 4. Pain will be recorded every 8 hours until discharge from the ICU, an average of 2 weeks, and at 6 months post discharge.
  Description of headache severity using headache scale score

SECONDARY OUTCOMES:
Opioid dose | 2 weeks (or duration of hospitalization)
  Amount of morphine equivalents/opioids used for pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binfalah M, Alghawi E, Shosha E, Alhilly A, Bakhiet M. Sphenopalatine Ganglion Block for the Treatment of Acute Migraine Headache. Pain Res Treat. 2018 May 7;2018:2516953. doi: 10.1155/2018/2516953. eCollection 2018. PMID 29862074
- [Background] Macdonald RL, Schweizer TA. Spontaneous subarachnoid haemorrhage. Lancet. 2017 Feb 11;389(10069):655-666. doi: 10.1016/S0140-6736(16)30668-7. Epub 2016 Sep 13. PMID 27637674
- [Background] Morad AH, Tamargo RJ, Gottschalk A. The Longitudinal Course of Pain and Analgesic Therapy Following Aneurysmal Subarachnoid Hemorrhage: A Cohort Study. Headache. 2016 Nov;56(10):1617-1625. doi: 10.1111/head.12908. Epub 2016 Oct 5. PMID 27704534
- [Background] Abraham MK, Chang WW. Subarachnoid Hemorrhage. Emerg Med Clin North Am. 2016 Nov;34(4):901-916. doi: 10.1016/j.emc.2016.06.011. PMID 27741994